CLINICAL TRIAL: NCT03293667
Title: Phenotypic and Functional Characterization of Regulatory T Lymphocytes in the Synovial Fluid of Patients Affected by Rheumatoid Arthritis, a Pilot Study.
Brief Title: Characterization of Regulatory T Lymphocytes in the Synovial Fluid of Patients Affected by Rheumatoid Arthritis.
Acronym: CATERLIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Default of recrutement / no more PI on this study
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL16_0264; 2016-A01489-42 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2017-03-16; First posted 2017-09-26 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis; Swelling Joint; Joint Fluid; Characterization of Regulatory T Lymphocytes
Keywords: Rheumatoid Arthritis; Regulatory T Cells
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exploratory arm (Other)
  Interventions: Other: Exploratory synovial fluid analysis

INTERVENTIONS:
Other: Exploratory synovial fluid analysis — An additional blood sample (3 10 ml tubes) and an additional specific analysis to characterize subpopulations of regulating T lymphocytes infiltrating the synovium of RA patients and comparing them with those of peripheral blood.

SUMMARY:
In rheumatoid arthritis (RA) the clinical response to anti-TNFα is related to an increase in the number or in the function of Treg lymphocytes in the peripheral blood of patients. This observation suggests the central role of Tregs in homeostasis of the immune response during RA.

In the literature the Tregs frequency and phenotype in the peripheral blood are well documented, however the analyses done on the Tregs in inflamed environment are still fragmentary or disparate.

In this project Tregs phenotype as well as expression of several transcripts will be analysed in order to better characterize the Treg cell subsets within the synovial fluid. Moreover, the local inflammatory cytokines (TNF, IL-6 and IL-1) may affect both the phenotype and the suppressive function of these Tregs and a comparison between peripheral and tissue Tregs will allow us to better understand the cause of functional loss.

Outcomes:

Primary outcome: Identification and characterization of the Tregs subpopulation present in the synovial fluid for RA patients suffering an episode of acute arthritis.

Secondary outcomes: compare the phenotypic and expression profile of the Tregs present in the synovial fluid with the Tregs present in the peripheral blood of RA patients suffering from an episode of acute arthritis.

DETAILED DESCRIPTION:
Transverse observational, monocentric exploratory study based on physiopathological evaluation Phase of identification/characterization of biomarkers. In a second phase, investigators might also considered a multicentre study with a greater number of patients as well as with osteoarthritis patients in order to validate the specificity of the results obtained in RA.

Investigators will prospectively recruit 10 patients with rheumatoid arthritis suffering from an episode of acute arthritis and requiring joint puncture. Investigators will analyse the cellular component of the joint fluid. It is an interventional clinical trial since one extra blood sample of 30 ml of blood will be collected.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* patients with rheumatoid arthritis according to 2010 ACR/EULAR criteria
* Patients with swelling joint suffering from an episode of acute articular flare link to RA and that requires an aspiration of joint fluid (RA with less than 3 months of evolution confirmed by clinical examination and/or joint ultrasound)
* Patients who agreed to participate to this study and signs the informed consent form

Exclusion Criteria:

* Septic arthritis confirmed by microbiological analysis of synovial fluid
* Osteoarthritis of the reference joint confirmed by X-ray
* Contraindication for joint aspiration: Platelets < 50 000/mm3, Prothrombin time <70%, Partial Thromboplastin Time Blood Test-PTT > 1,5 times compare to the control sample, anticoagulant therapy
* Biotherapy (including (anti-TNF-α), corticosteroid (orally, intravenously or intra-articulary) or others immunosuppressive drug (current treatment or treatment within 3 months before joint aspiration).
* Pregnancy, mother in the post natal period or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Define the heterogeneity of Treg cell subsets | Through study completion, an average of 2 years
  Description of Treg cell subsets isolated from the synovial fluid of RA patients suffering from an episode of acute arthritis.

SECONDARY OUTCOMES:
Compare the phenotypic and expression profile of the Tregs | Through study completion, an average of 2 years
  Comparison between the phenotypic and expression profile of the Tregs present in the synovial fluid with the Tregs present in the peripheral blood of RA patients suffering from an episode of acute arthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- Lapeyronie Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No